CLINICAL TRIAL: NCT03409445
Title: Validation of a Food Frequency Questionnaire for the Assessment of Omega-3
Brief Title: Validation of a Food Frequency Questionnaire for the Assessment of Omega-3 Fatty Acid Intake
Status: Completed | Type: Observational
Sponsor: Isabelle Herter-Aeberli (Other)
Collaborators: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, Principle investigator, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Other Study IDs: N3FFQ
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention (observational study)

SUMMARY:
As essential nutrients omega 3 fatty acids contribute to normal growth and development. Inadequate intake is linked to the development of chronic diseases such as coronary heart disease, high blood pressure, cancer, arthritis, psychological illnesses and allergies. Therefore, it is important to be able to reliably detect the intake of these fatty acids. Due to eating habits varying in different countries the questionnaire documenting dietary habits needs to be adapted to the situation in question. Based on a US version the investigators developed a questionnaire suitable for Switzerland and now wish to validate it by measuring the fatty acid composition of red blood cells, which will provide information on the intake of the various fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females aged 18 to 60

Exclusion Criteria:

* known disorders of the gastrointestinal tract which can lead to malabsorption
* intake of medication which could affect the absorption of any nutrients
* Pregnant or breast-feeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Fatty acid composition of red blood cells due to dietary habits | 1 day ( first visit)
  Fatty acid composition of red blood cells due to dietary habits

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Switzerland